CLINICAL TRIAL: NCT05758246
Title: Senolytics To slOw Progression of Sepsis (STOP-Sepsis) Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRP-XXX
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; Acute Infection; Organ Failure
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Participants will initially be equally randomized between placebo, 20 mg/kg (once), and 20 mg/kg (once daily for 2 days). After 60 participants have been enrolled, the randomization ratio will be adapted so that a higher proportion of participants will be randomized to the optimal dosing regimen. The proportion randomized to the control will be held constant throughout the trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fisetin- dose 1 (Experimental): Elderly (>=65 years) patients admitted to the hospital with an acute infection and sequential organ failure assessment score sufficient for a diagnosis of sepsis, will be given the first dose of fisetin.
  Interventions: Drug: Fisetin-dose 1
- Fisetin- dose 2 (Experimental): Elderly (>=65 years) patients admitted to the hospital with an acute infection and sequential organ failure assessment score sufficient for a diagnosis of sepsis, will be given the 2nd does of fisetin.
  Interventions: Drug: Fisetin-dose 2
- Placebo (Placebo Comparator): Elderly (>=65 years) patients admitted to the hospital with an acute infection and sequential organ failure assessment score sufficient for a diagnosis of sepsis will receive placebo treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin-dose 1 — 20mg/kg once a day for one day.
  Arms: Fisetin- dose 1
Drug: Fisetin-dose 2 — 20mg/kg once a day for two days
  Arms: Fisetin- dose 2
Drug: Placebo — Placebo treatment
  Arms: Placebo

SUMMARY:
The long-term goal is to test the clinical efficacy of senolytic therapies to reduce progression to and severity of sepsis in older patients. The central hypothesis is that a threshold burden of SnCs predisposes to a SASP mediated dysfunctional response to PAMPs, contributing to a disproportionate burden of sepsis in older patients. The study hypothesizes timely treatment with fisetin will interrupt this pathway.

A multicenter, randomized, adaptive allocation clinical trial to identify the most efficacious dose of the senolytic fisetin to reduce the composite cardiovascular, respiratory, and renal sequential organ failure assessment score at 1 week, and predict the probability of success of a definitive phase III clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age >=65 years
* Primary diagnosis of acute infection (per investigator judgment)
* SOFA >1
* Admission order to the hospital
* Expected length of stay >=48 hours (per investigator judgment)

Exclusion Criteria:

* Admission to the ICU
* Vasopressors, mechanical ventilation, or dialysis
* Comfort care only
* Total bilirubin >3X or AST/ALT >4x upper limit of normal
* eGFR < 25 ml/ min/ 1.73 m2
* Hemoglobin <7 g/dL; white blood cell count ≤ 2,000/mm3; absolute neutrophil count ≤1 x 10^9/;, or platelet count ≤ 40,000/μL
* Known HIV, Hepatitis B, or Hepatitis C
* Invasive fungal infection (per investigator judgment)
* Uncontrolled effusions or ascites (per investigator judgment)
* New/active invasive cancer except non-melanoma skin cancers
* Known hypersensitivity or allergy to Fisetin.
* Active treatment with potential drug-drug interactions
* Enrolled in another sepsis clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-08-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Difference in the composite cardiovascular, respiratory, and renal sequential organ failure assessment (CRR-SOFA) | day 7
  The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category. This outcome assesses only the cardiovascular, respiratory, and renal categories of the total SOFA score, and calculates the change from day 0 to day 7.

SECONDARY OUTCOMES:
Safety of 2 doses of fisetin in patients with mild sepsis | day 28
  Outcome is the number of serious adverse event
Organ failure free days | day 28
  Outcome is 28 days minus the last day the patient required any of the following: ventilator support, vasopressors, or dialysis / renal replacement therapy. Patients who die prior to day 28 are given a value of -1.
Total SOFA score | day 7
  The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category.
Zubrod performance status | day 7
  A scale for indicating a patient's functional level: 0 asymptomatic - 1 Symptomatic, fully ambulatory - 2 Symptomatic, in bed - 50% of the day - 3 Symptomatic, in bed; 50% of the day but not bedridden - 4 Bedridden - 5 Dead.
SF-12 score | day 7
  The SF-12 is a self-reported validated outcome measure assessing the impact of health on an individual 39;s everyday life. Patients fill out a 12 question survey which is then scored by a clinician or researcher.
SF-12 score | day 28
  The SF-12 is a self-reported validated outcome measure assessing the impact of health on an individual 39;s everyday life. Patients fill out a 12 question survey which is then scored by a clinician or researcher.
Zubrod performance status | day 28
  A scale for indicating a patient's functional level: 0 asymptomatic - 1 Symptomatic, fully ambulatory - 2 Symptomatic, in bed - 50% of the day - 3 Symptomatic, in bed; 50% of the day but not bedridden - 4 Bedridden - 5 Dead.
Days in the ICU | day 28
  This outcome is the number of days the patient was admitted to the ICU.
All-cause mortality | Day 28
  This outcome is the proportion of patients suffering all-cause mortality prior to day 28.
Peripheral CD3+ senescent (SnCs) immune cells | day 7
  Outcome is the relative expression of p16Ink4a in CD3+ cells.
Outcome is the relative expression of p16Ink4a in CD3+ cells. | day 28
  Outcome is the relative expression of p16Ink4a in CD3+ cells.
TNF-alpha | day 7
  Outcome is the concentration of TNF-alpha by Luminex human discovery assay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Puskarich, MD, Principal Investigator — University of Minnesota
Locations (10):
- United States (10):
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Ridges, Burnsville, Minnesota
  - Southdale, Edina, Minnesota
  - M Health Fairview St. John's, Maplewood, Minnesota
  - St. John's, Maplewood, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - HCMC, Minneapolis, Minnesota
  - UMMC, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva M, Wacker DA, Driver BE, Staugaitis A, Niedernhofer LJ, Schmidt EL, Kirkland JL, Tchkonia T, Evans T, Serrano CH, Ventz S, Koopmeiners JS, Puskarich MA; STOP-Sepsis Investigators. Senolytics To slOw Progression of Sepsis (STOP-Sepsis) in elderly patients: Study protocol for a multicenter, randomized, adaptive allocation clinical trial. Trials. 2024 Oct 21;25(1):698. doi: 10.1186/s13063-024-08474-2. PMID 39434114